CLINICAL TRIAL: NCT05126420
Title: A RARE TUMOR OF THE ORAL MUCOSE, MIYOPERİCYTOMA: CASE REPORT
Brief Title: MIYOPERİCYTOMA OF ORAL MUCOSE: CASE REPORT
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Elif Polat, research assistant, Ankara University
Other Study IDs: elıfpolat
Record Dates: First submitted 2021-10-04; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Myopericytoma
Keywords: oral pathology; mıyopericytoma
MeSH Terms: conditions — Myopericytoma | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — A sample was taken from the lingual region of the mandible for pathology.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: biopsy — biopsy to identify the lesion in the oral mucosa

SUMMARY:
Miyopericytoma (MPC) is defined as a benign tumor consisting mostly of oval-spindle-shaped myoid-appearing cells with perivascular growth. It may involve a single or multiple anatomical regions and may be multifocal and tends to occur mainly in the extremities, dermal and superficial soft tissues of adults. Cases of miyopericytoma due to trauma have been reported.Histological features and clinical course are generally benign, but features suggestive of low-grade malignancy were seen in MPCs. Myopericytoma in the oral and maxillofacial region is rare and a limited number of cases have been reported in the literature.

A 42-year-old female patient was admitted to our clinic with an enlarging lesion on the lingual aspect of the anterior mandible, which she noticed 2 years ago. As a result of the examination, a smooth-surfaced, off-white, pedunculated, fibrotic, painless, and non-bleeding lesion was detected in the lingual aspect of the anterior mandible. The lesion was removed by excisional biopsy.

ELIGIBILITY:
Inclusion Criteria:

Patient with a fibrotic lesion in the mouth

Exclusion Criteria:

Patient without fibrotic lesions in the mouth.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
biopsy | 2 day
  We evaluated the extracted biopsy material with histological parameter.

SECONDARY OUTCOMES:
recurrence | 1 year
  Clinical parameter

CONTACTS AND LOCATIONS:
Overall Officials: elif polat, Principal Investigator — dtelifpolat@gmail.com
Locations (1):
- Elif Polat, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided